CLINICAL TRIAL: NCT03177772
Title: Group Therapy For Dementia Caregivers At Risk For Complicated Grief
Acronym: PLGT
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Principal Investigator, Katherine Supiano, Associate Professor, University of Utah
Other Study IDs: AARG-17-503706
Record Dates: First submitted 2017-05-26; First posted 2017-06-06 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Grief
Keywords: caregivers; grief; dementia; long-term care; psychotherapy group
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- LTC Facility 1: Pre-loss Grief Support Group offered in long-term care facility for dementia family caregivers anticipating the death of their care recipient within next 6 month. Two hour sessions for 10 weeks include psychoeducation, motivational interviewing, cognitive behavioral and exposure approaches. Supportive others, selected by participants are included in two sessions.
  Interventions: Behavioral: Pre-loss group therapy
- LTC Facility 2: Pre-loss Grief Support Group offered in long-term care facility for dementia family caregivers anticipating the death of their care recipient within next 6 month. Two hour sessions for 10 weeks include psychoeducation, motivational interviewing, cognitive behavioral and exposure approaches. Supportive others, selected by participants are included in two sessions.
  Interventions: Behavioral: Pre-loss group therapy
- LTC Facility 3: Pre-loss Grief Support Group offered in long-term care facility for dementia family caregivers anticipating the death of their care recipient within next 6 month. Two hour sessions for 10 weeks include psychoeducation, motivational interviewing, cognitive behavioral and exposure approaches. Supportive others, selected by participants are included in two sessions.
  Interventions: Behavioral: Pre-loss group therapy

INTERVENTIONS:
Behavioral: Pre-loss group therapy — The PLGT intervention will include CGGT treatment elements modified to address the pre-loss preparation of caregivers at risk for complicated grief, and will focus on the perceived relationship and attachment status between caregiver and care recipient, how memories of the life together, the illness and the death are interpreted, and strategies for preparing for life without the care recipient. These activities include elements of motivational interviewing, cognitive behavioral therapy and prolonged exposure therapy.

SUMMARY:
The investigators are adapting Complicated Grief Group Therapy (CGGT) for soon-to-be bereaved dementia caregivers at risk for complicated grief-Pre-Loss Group Therapy (PLGT) to facilitate healthy death preparedness and eventual bereavement. This will be the first known application of proven therapeutic strategies to address complicated grief applied to high-risk dementia caregivers prior to care recipient death to mitigate complicated grief. If proven to be effective in attenuating poor bereavement outcomes, PLGT could be translated into comprehensive caregiver support programs and delivered to active caregivers of living persons with dementia at risk for complicated grief through community-based caregiver support groups.

DETAILED DESCRIPTION:
In the investigators previous evaluation of Complicated Grief Group Therapy (CGGT) in bereaved dementia caregivers (2014-NIRG-305569), CGGT was administered to participants in a prospective, randomized-controlled trial. Participants in 5 treatment groups confirmed clinically significant reduction in complicated grief on the Inventory of Complicated Grief. In that study, intervention elements suitable for adaption in a preventative care approach were identified. The investigators are adapting these elements of CGGT for soon-to-be bereaved dementia caregivers at risk for complicated grief-Pre-Loss Group Therapy (PLGT) to facilitate healthy death preparedness and eventual bereavement.

Specific Aims: 1) Assess preparedness for death and grief of bereaved and soon-to-be bereaved caregivers. 2) Adapt CGGT treatment elements into a manualized pre-loss preparedness group psychotherapy-(PLGT)-for dementia caregivers at risk for complicated grief. 3) Implement and evaluate three PLGT cohorts (NTotal = 40) in three long-term care facilities with family caregivers at-risk for complicated grief whose care recipient has a life expectancy of 6 months or less and resides in a long-term care facility.

ELIGIBILITY:
Inclusion Criteria:

* Study participants will be ADRD caregivers at risk for CG with a family member diagnosed with ADRD having a life expectancy of less than 6 months and residing in the facility. Caregivers with ADRD residents nearing death will be temporally closer to their grief/preparedness experience permitting 3 month post death follow-up within the study timeline. Eligibility (stage 1). Potential family caregiver participants will be identified by facility leadership (Medical Director, Social Worker and Director of Nursing) by these inclusion criteria:

  1. resident ADRD diagnosis,
  2. life expectancy, "Would you be surprised if this resident died in the next 6 months?" and
  3. caregiver proximity to facility permitting participation. Potential participants will receive an invitation phone call from the ResearchAssistant (RA). Eligibility (stage 2). Interested individuals will be invited to a pre-screening interview with the RA in person at the facility. Those who meet the final inclusion criteria,
  4. minimum score of 4 on p-BGQ, and
  5. positive scores on 4 of 9 risk factors will qualify

Exclusion Criteria:

* Active suicidality (likely hospitalization) will exclude interested individuals from participating

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study participants will be ADRD caregivers at risk for CG with a family member diagnosed with ADRD having a life expectancy of less than 6 months and residing in one of three partner Long-term care the facilities
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Grief | 3 months post death of care recipient
  Change in pre-loss grief as measured by Inventory of Complicated Grief-revised (Prigerson, et al., 1995; ICG-r)

SECONDARY OUTCOMES:
Meaning Making | 3 months post death of care recipient
  Change in meaning making as measured by Grief and Meaning Reconstruction Inventory, (Gillies, et al., 2015; GMRI)
Preparedness | 3 months post death of care recipient
  Change in perceived preparedness for death of care recipient as measured by Preparedness question; "How prepared are you/were you for the death of your (spouse/parent)?" (Herbert, Dang & Schulz, 2006).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - St. Joseph Villa, Salt Lake City, Utah
  - Silverado Care Facility, Salt Lake City, Utah
  - William E. Christoffersen Veterans Home, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided
Research protocol is registered in Open Science Framework. Individual de-identified participant data available only through direct request to PI.

REFERENCES:
- Available data/document: Study Protocol: dtp38 — https://osf.io/dtp38/ — Open Science Framework. we are registered